CLINICAL TRIAL: NCT02571413
Title: Evaluation of the Animated Cartoon-aided Teaching of Intranasal Corticosteroid Administration Technique Among Thai Children With Allergic Rhinitis
Brief Title: Evaluation of the Animated Cartoon-aided Teaching of Intranasal Corticosteroid Allergic Rhinitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nualanong Visitsunthorn (Other)
Collaborators: Siriraj Hospital (Other)
Responsible Party: Sponsor-Investigator, Nualanong Visitsunthorn, Somying Indradat, Mahidol University
Organization: Mahidol University (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: [Si 9091/2552(EC2)]
Record Dates: First submitted 2010-01-11; First posted 2015-10-08 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Asthma; Allergic Rhinitis
Keywords: animated cartoon-aided teaching; oral presentation; allergic rhinitis; intranasal corticosteroid; how to use intranasal corticosteroid
MeSH Terms: conditions — Asthma; Rhinitis, Allergic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- oral presentation (Other): Scoring the correct use of INC before, immediate after and 3 months after oral presentation without demonstration "how to use INCS"
  Interventions: Other: score before teaching; Other: score immediately after teaching; Other: score 3 months after teaching
- animated cartoon-aided VDO (Other): Scoring the correct use of INC before, immediate after and 3 months after animated cartoon-aided teaching "how to use INCS"
  Interventions: Other: score before teaching; Other: score immediately after teaching; Other: score 3 months after teaching

INTERVENTIONS:
Other: score before teaching — score the check-point of correct INCS usage before teaching
Other: score immediately after teaching — score the check-point of correct INCS usage immediately after teaching
Other: score 3 months after teaching — score the check-point of correct INCS usage 3 months after teaching

SUMMARY:
Correct methods and compliance of intranasal corticosteroid (INCS) is very important for the treatment of allergic rhinitis (AR). The animated cartoon-aided teaching of INCS administration was created to decrease workload of health care professionals. The aim of this study is to compare the achievement of the children with AR in using INCS between the group which were instructed by animated cartoon-aided teaching or oral presentation without demonstration.

DETAILED DESCRIPTION:
The study was a prospective randomized control trial in children aged 5 - 16 years with moderate to severe intermittent or persistent AR who had never used INCS. The patients were randomly divided into 2 groups; 1) Teaching how to use INCS by oral presentation and 2) by animated cartoon-aided teaching. Successful achievements were recorded when the patients were able to use INCS (all five-point checklists) correctly. If they were unable to use the INCS correctly after the first teaching, the same instruction would be repeated and the second assessment would be performed.

ELIGIBILITY:
Inclusion Criteria:

* Children with 5 - 16 year old
* children with allergic rhinitis

Exclusion Criteria:

* history of intranasal corticosteroid use
* history of other underlying disease

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2009-05; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Scores of the correct method of intranasal corticosteroid administration technique before and after teaching | 1 year
  compare the scores before and after teaching( immediately and 3 months after)

CONTACTS AND LOCATIONS:
Overall Officials: Nualanong Visitsunthorn, Prof, Principal Investigator — Mahidol University
Locations (1):
- Siriraj hospital, Mahidol University, Bangkok, Bangkok, Thailand